CLINICAL TRIAL: NCT01549080
Title: A Double-blind, Placebo-controlled, Randomized, Parallel-group Study of the Safety and Effects of YisuiShengxueGranules on Thalassemia Presenting the Syndrome of Deficiency of Liver/Kidney-yin, and Asthenia of Essence/Blood.
Brief Title: Study of Effects of YisuiShengxueGranules on Thalassemia
Acronym: thalessemia
Status: Completed | Type: Observational
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Wu Zhikui，Prof., Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Other Study IDs: 2011001P02/June 3rd, 2011; 2010CB530406 (Other Grant/Funding Number: Ministry of science and technology "973" project)
Record Dates: First submitted 2012-02-27; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2011-06

CONDITIONS: Thalassemia
Keywords: traditional chinese medicine and thalassemia
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood and bone marrow cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- research: biological research on the effects of yisuishengxuegranule
  Interventions: Drug: Yisuishengxue Granule
- clinical research: clinical research on thalassemia
  Interventions: Drug: Yisuishengxue Granule

INTERVENTIONS:
Drug: Yisuishengxue Granule — Yisui Shengxue Granules，produced by pharmaceutical factory of Guang'anmen Hospital, China Academy of Chinese Medical Sciences, is made from the herbs of Shan Zhu Yu (Fructus Corni), He Shou Wu (Radix Polygoni Multiflori), Shu Di Huang (Radix Rehmanniae Preparata), Huang Qi (Radix Astragali) and etc.Yisui Shengxue Granules：12g/bag， Registration Number：20110602； Yisui Shengxue Granules replacer (placebo)：12g/bag，Registration Number：20110519；Treatment group：Yisui Shengxue Granules，1 bag, tid, po； Control group: Yisui Shengxue Granules replacer (placebo), 1 bag, tid, po; Intervention for 12 weeks. Follow-up 3 months later after stopping the drug intervention.
  Other Names: Yisui Shengxue Granules replacer (placebo)：

SUMMARY:
The primary objectives of this study are to evaluate whether Yisui Shengxue Granules therapy can increase the hemoglobin level in peripheral blood and alleviate the symptoms, and at the same time, evaluate its safety in the treatment of Thalassemia with the syndrome of deficiency of liver-yin and kidney-yin, and asthenia of essence and blood.

DETAILED DESCRIPTION:
3. INVESTIGATION PLAN 3.1 Study Design and Plan This study is a double-blind, placebo-controlled, randomized Parallel-group trial. Guang'anmen Hospital is the sponsor and has designed the clinical trial protocol. No.303 Hospital of Chinese People's Liberation Army (PLA) is the collaborator, where the most patients come from.

3.2 Random Method Using the randomized block design，stratifying by α-Thalassemia and β-Thalassemia, the patients will be allocated randomly 1:1 to Yisui Shengxue Granules group or placebo group.

Statistic Analysis System (SAS, SAS institute, Cary, NC, USA) was used to produce 001~120 random code, matching 120 subjects who divided randomly 1:1 into Yisui Shengxue Granules group and placebo group.

3.3 Blinding Design 3.3.1 Packaging of the study drug and placebo: all drugs including medical emergency envelops must be repackaged and reallocated according to regulations of standard double-blind clinical trial.

3.3.2．Blinding The encoded data will be kept in Guang'anmen Hospital, China Academy of Chinese Medical Sciences.

When all patients fulfill the procedures of the trial, the data will be entered into electronic Case Report Forms (eCRFs) and locked, and then the blind will be disclosed.

If unmasking is necessary because of a serious, unexpected and related adverse event or if a medical emergency occurs which requires knowledge of the exact therapy, the investigator may contact the principal investigator or censor to determine whether the medical emergency envelop will be broken. The date and reason of the code breaking must be documented and signed and this information must be sent to the sponsor and collaborator. The patient should be withdrawn from Study Medication but be followed up according to the protocol.

If twenty percent medical emergency envelops are broken or blinding method is betrayed, this trial will be fail.

3.4 Sample Size Estimation A total of 120 patients will be required (α-Thalassemia: 80, β-Thalassemia: 40 ), assuming a relative risk of sample loss (no more than 20%) in the whole trial-- an accrual period of 3 months treatment and a minimum 3 months follow up. The numbers of patients in both study drug group and placebo group are equal.

4.6 Removal of Patients from Study 4.6.1 Investigators make the decision of patients' withdrawal.

Investigators will decide to withdraw the patients if they have following conditions in the middle of the trial:

1. Upper respiratory tract infection with temperature higher than 38.5℃. This condition will lead to hemolysis aggravation and hemoglobin level decreasing, affecting the evaluation of therapeutic effects. The patients will be regarded as invalid cases once they withdraw from the trial and accept other therapy.
2. Anemia complications or physiological changes make the patients being unsuitable to continue in this clinical study.
3. Patients, with poor compliance, take the Study Medication less than 80% or more than 120%.
4. Unblinding cases and unmasking cases because of medical emergency.
5. Taking prohibited drugs.
6. Refusing to take any Study Medication. 4.6.2 Patients make the decision of their withdrawal. In accordance with the World Medical Association Declaration of Helsinki (1996 version), as amended from time to time, all patients have the right to withdraw from the study at any time and for any reason, without prejudice to his or her future medical care by the physician or institution, and is not obliged to give his or her reasons for doing so. Without compromising the right of patients to withdraw from the trial, every effort will be made to understand and accommodate their concerns and avoid withdrawal wherever possible. If patients do not fulfill the therapy, tests, or follow-up for any reason, the patients will be dealt with as removal from the study.

4.6.3 The case report forms of withdrawal patients, for whatever reason, must be kept. The last test results will be dealt with as the terminal results to enter the full analysis set. If the significant effects are showed up in less than 3 moths, the patients will be considered as significant effective cases though they complete the trial in advance.

4.7 Termination Criteria Trial termination means the study may be terminated at any time if the study represents a serious medical risk to the patients.

1. Serious safety risk.
2. Gross error in the clinical trial protocol or major deviation appears during trial execution.
3. Sponsor's request (reasons of finance, administration, etc.)

5.3 The Packaging Boxes and Preservation In a large packaging box, there will be three medium size packing boxes, containing 3 months dosage of Study Medication for one patient. The Study Medication can be either Yisui Shengxue Granules or placebo according to the random code, preserved by specially-assigned person and stored in dry environment at room temperature.

5.4 Drugs Assignment, Checking and Return Study Medication will be delivered to each clinical center according to the Study Medication code that randomly assigned to the clinical center, and be distributed to patients, who fulfill the inclusion criteria, in the order of drug code in 3 times. "Drug Used Report" should be filled in timely and kept by drug administrator.

Investigators should record the Study Medication quantity that patients received, took, and returned when they visit.

5.5 Drugs Blinding and Medical Emergency Envelope Study Medication blinding will be made by the corresponding department according to the randomization list. A medical emergency envelope, with detailed information of the medication, will be prepared for every randomization code and be kept in the principal investigator of each clinical center.

5.6 Precautions and Prohibited Drug Combination

1. In this Trial, other drugs for β-Thalassemia are prohibited.
2. Patients, taking other drugs for other diseases, should be recorded in the item "the table for being using other drugs for other diseases" in CRF.

6. OBSERVATIONS AND MEASUREMENTS 6.1 General Conditions (Before Entering the Trial)

1. Record age, gender, body weight and height.
2. Record past medical history: course of disease, diagnosis by Western Medicine and Chinese Medicine, type of Thalassemia, course of treatment, combined diseases and concomitant medication.

6.2 Indexes for Safety Evaluation (Before and After the Trial)

(1) Temperature, blood pressure, respiratory rate and heart rate (2) Routine tests of blood, urine and stool (3) ECG (4) Liver function (ALT) (5) Kidney function (BUN, Cr) (6) Record any relevant adverse events 6.3 Indexes for Therapeutic Effects Evaluation 6.3.1 Major indexes

1. Clinical effects: screening visit (visit 1), visit 2 (4 weeks later), visit 3 (8 weeks later), visit 4 (12 weeks later, the end of the medication therapy), visit 5 (follow-up 3 months later after medication therapy).
2. Chinese Medicine syndrome improvment: screening visit (visit 1), visit 2 (4weeks later), visit 3 (8 weeks later), visit 4 (12 weeks later, the end of the medication therapy), visit 5 (follow-up 3 months later after medication therapy).

6.3.2 Secondary indexes

1. Blood tests: white blood cell, hemoglobin, red blood cell, reticulocyte percentage, hemoglobin eletrophoresis, fetal Hb, HbA2, HbH, platelet. Screening visit (visit 1), visit 2 (4weeks later), visit 3 (8 weeks later), visit 4 (12 weeks later, the end of the medication therapy), visit 5 (follow-up 3 months later after medication therapy).
2. Hepatic oblique diameter and spleen horizontal diameter by ultrasound imaging test (Before and after trial).
3. Improvement of individual symptom: Screening visit (visit 1), visit 2 (4weeks later), visit 3 (8 weeks later), visit 4 (12 weeks later, the end of the medication therapy), visit 5 (follow-up 3 months later after medication therapy).

8. ADVERSE EVENTS 8.1 Adverse Event Record During the trial, if adverse events happen, the occurrence time, severity, duration, therapeutic measures and clinical outcomes must be recorded authentically in "DRUG ADVERSE EVENT FORM".

8.2 Severity of the Adverse Event

The severity of adverse events should be graded as follows:

Mild: Mild, tolerable discomfort, no need for special management, no influence to the trial and patient's rehabilitation.

Moderate: Moderate and intolerable discomfort, special management is necessary, having direct influence to patient's rehabilitation.

Severe: Severe discomfort, life-threatening, death or disability is possible and emergency intervention is necessary.

8.3 Relationship to Study Medication 8.3.1 Identification standards

1. Whether there is a reasonable relationship between the time of taking Study Medication and the occurrence of the suspected adverse reactions.
2. Whether the suspected adverse reactions accord with the adverse reactions known to the Study Medication.
3. Whether the suspected adverse reactions can be interpreted as the results of drugs combination, patient's clinical condition, or other therapies.
4. Whether the suspected adverse reactions disappear or are relieved by reducing the Study Medication dosage or stopping to take.
5. Whether the suspected adverse reactions occur again at the time of retaking the suspected drugs? Adverse Reaction Identification Conclusions Items 1 2 3 4 5 Sure + + - + + Probable + + - + ？ Undetermined + + ± ± ？ Unlikely + - ± ± ？ Unconcerned - - + - - Note：+ Yes, - No, ± uncertain, ？Information is not available 8.3.2 According to the above table, the relationship between adverse reaction and Study Medication will be classified into 5 kinds as following: 1-sure, 2-probable, 3-undetermined, 4-unlikely 5-unconcerned The incidence rate of adverse reactions =（the number of cases with adverse reactions including kind 1, 2 and 3）/（the number of cases which need to be identified whether adverse reactions happen） 8.4 Adverse Event Handling 8.4.1 Handling principle：Any adverse events such as patients' complaints and laboratory abnormality should be taken seriously and analyzed carefully. Measures for managing adverse reactions should be taken at once to protect the patients.

8.4.2 Handling Procedure：Adverse reactions should be documented in CRF in detail including rechecking (when it is necessary), duration, prognosis and relief.

8.4.3 Serious Adverse Events Handling

1. During the Trial, any serious adverse events must be reported to the clinical center, sponsor and medical ethics committee and recorded in "DRUG ADVERSE EVENT FORM". All clinical centers, principal investigators and the contact person listed on the CFR should be informed as well at same time. Besides, a serious adverse reaction must be reported to the State Food and Drug Administration within 24 hours.
2. Measures：If a medical emergency happens to a patient, the corresponding medical emergency envelop will be broken by the principal investigator of the clinical center in the presence of two witnesses. Proper management for adverse reactions will be taken and CRA should be informed the outcomes. Investigators should write down the information including unblinding reason, date, management and outcomes in CRF and sign their names.

8.4.4 Following up Adverse Events Unrelieved Any adverse events should be followed up until the adverse reactions relief or being stable.

ELIGIBILITY:
Inclusion Criteria:

1. Intermedia α-Thalassemia; intermedia β-Thalassemia; severe β-Thalassemia.
2. Syndrome of Deficiency of Liver-yin and Kidney-yin, and Asthenia of Essence and Blood.
3. Male or female, 3-40 years of age.
4. Provision of written informed consent.

Exclusion Criteria:

1. Complications with critical illness such as cerebrovascular disease, cardiovascular disease, hepatic disease, renal disease, malignancy and etc.
2. Allergy to any ingredients of Yisui Shengxue Granules
3. Psychiatric disorder.
4. Blood transfusion in the latest 90 days for severe β-Thalassemia; blood transfusion in the latest 45 days for intermediaβ-Thalassemia or intermedia α-Thalassemia.。
5. Upper respiratory tract infection with temperature higher than 38.5℃ in the latest 45 days.
6. Taking other antianemic agents in the latest 2 months.
7. Participation in any other clinical interventional trial in the latest 1 month.

Ages: 3 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The type of severe β-Thalassemia：Hb <60g/L, microcytic hypochromic anemia; more than 10% target erythrocyte and erythrocyte fragments; increased number of reticulocyte; more erythroblast in peripheral blood; extremely proliferative in marrow; HbF>30%～90%.
  The type of intermedia β-Thalassemia：Hb 60g/L～100g/L; the shape of mature erythrocyte is similar to severe type; more reticulocyte; erythroblast may be found; HbF>3.5%.
  The type of intermedia α-Thalassemia： The patients have mild or moderate anemia (Hemoglobin in a few patients is less than 60g/L or more than 100g/L)，probably have hepatosplenomegaly, jaundice, and Mediterranean anemia features.
  The Diagnosing Criteria for the Deficiency Syndrome of Liver-yin and Kidney-yin, and Asthenia of Essence and Blood in Chinese Medicine
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Clinical effects on heamoglobin changes | 6 months
  Changes from Baseline in heamoglobins at 3and 6 months

SECONDARY OUTCOMES:
Chinese Medicine syndrome improvment | 6 months
  changes from baseline in syndromes at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wu zhikui, MD, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences

REFERENCES:
- [Derived] Foong WC, Loh CK, Ho JJ, Lau DS. Foetal haemoglobin inducers for reducing blood transfusion in non-transfusion-dependent beta-thalassaemias. Cochrane Database Syst Rev. 2023 Jan 13;1(1):CD013767. doi: 10.1002/14651858.CD013767.pub2. PMID 36637054
- [Derived] Cheng YL, Zhang XH, Sun YW, Wang WJ, Huang J, Chu NL, Fang SP, Wu ZK. Genomewide DNA Methylation Responses in Patients with beta-Thalassemia Treated with Yisui Shengxue Granules (). Chin J Integr Med. 2019 Jul;25(7):490-496. doi: 10.1007/s11655-018-2777-9. Epub 2018 May 3. PMID 29761313